CLINICAL TRIAL: NCT03414632
Title: Prevalence of Transthyretin Cardiac Amyloidosis in Heart Failure With Preserved Ejection Fraction: A Community Study
Brief Title: Transthyretin Cardiac Amyloidosis in HFpEF
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Omar Abou Ezzeddine, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-003021
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; Diastolic Heart Failure; Heart Failure with Preserved Ejection Fraction; Transthyretin Cardiac Amyloidosis; Amyloidosis
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic; Amyloidosis | interventions — Technetium Tc 99m Pyrophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPECT/CT (Other): 99mTc-PYP single-photon positive emission computed tomography with computed tomography
  Interventions: Drug: 99mTc-PYP

INTERVENTIONS:
Drug: 99mTc-PYP — Radioisotope used in the SPECT/CT imaging

SUMMARY:
To estimate the prevalence of transthyretin cardiac amyloidosis (TTR-CA) among Heart Failure with Preserved Ejection Fraction (HFpEF) patients with increased LV wall thickness in Southeast Minnesota using 99mTc-PYP single-photon positive emission computed tomography with computed tomography (SPECT/CT).

DETAILED DESCRIPTION:
Residents of Southeast Minnesota over 60 years of age with an inpatient or outpatient diagnosis of heart failure (HF) will be consecutively identified in real-time using a natural language processing (NLP) search engine, their HF diagnosis validated, and those with a recent (≤ 12 months) echocardiogram documenting a preserved EF( ≥ 40%) and LV wall thickening will be consented to undergo venipuncture, urine collection and 99mTc-PYP SPECT/CT imaging to rule in/out the diagnosis of TTR-CA. Hence, the prevalence of TTR-CA will be defined. To place this prevalence in perspective of the global HFpEF cohort in the community, a rigorous screening log will be maintained to allow generation of a comprehensive CONSORT diagram. Importantly, baseline characteristics of patients who qualify for our study but decline to consent will still be collected provided that consent for use of their records for medical research had previously been granted.

ELIGIBILITY:
Inclusion Criteria

1. Resident of Southeastern Minnesota (Olmsted, Dodge, Fillmore, Mower, Freeborn, Wabasha, or Steele County)
2. Current diagnosis of HF per NLP search
3. Age > 60 years
4. Clinically obtained echocardiogram within 12 months of index visit showing:

   1. EF ≥ 40% and
   2. Increased Left Ventricular (LV) wall thickness as defined by an end-diastolic left ventricular septal or posterior wall thickness (LVWTd) ≥ 20% above the upper limit of normal measured by 2D or M-mode imaging in the parasternal long (2D) or short (M-mode) axis view (≥12 mm).
5. Objective evidence of HF defined as one or more of the following present within 24 months of index visit:

   1. Meet Framingham Criteria at index visit (In-patient or outpatient)
   2. Previous HF hospitalization
   3. Invasive hemodynamic documentation of elevated pulmonary capillary wedge pressure (PCWP) or left ventricular end-diastolic pressure (LVEDP) (> 18 mmHg at rest or > 25 mmHg with exercise)
   4. Left atrial enlargement + loop diuretic for HF(clinically obtained) N-terminal pro b-type natriuretic peptide (NT-proBNP) > 300 (sinus rhythm) or >900 (atrial fibrillation) pg/mL

Exclusion Criteria

1. Documentation of previous EF < 40%
2. Any cardiac surgery or major chest trauma within 4 weeks of index visit
3. Presence or history of hemodynamically significant left sided valvular disease defined as:

   1. Greater than mild mitral stenosis
   2. Intrinsic mitral valve disease (prolapse, flail) with greater than moderate regurgitation
4. Myocardial infarction within 4 weeks of index visit defined by typical angina, EKG changes and significant change in serial troponins. Note that chronic troponin elevation is extremely common in cardiac amyloidosis. Hospitalized patients with troponin elevation but no significant change (delta) on serial testing will NOT be excluded.
5. Prior or current exposure to Plaquenil (Hydroxychloroquine)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of TTR-CA | Baseline
  Determine the prevalence of Transthyretin Cardiac Amyloidosis in a community based cohort of consecutive Heart Failure with Preserved Ejection Fraction patients with increased Left Ventricular wall thickness using 99mTc-Pyrophosphate (99mTc-PYP) single-photon positive emission computed tomography with computed tomography (SPECT/CT).

CONTACTS AND LOCATIONS:
Overall Officials: Omar F Abou Ezzeddine, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials